CLINICAL TRIAL: NCT05436184
Title: Influenza IMPRINT Cohort: Defining the Impact of Initial Influenza Exposure on Immunity in Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1U01AI144673-01 (NIH); 1U01AI144673-01 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Influenza
Keywords: influenza, birth cohort
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs will be obtained weekly and will be tested for influenza A & B viruses by Real-Time Reverse Transcriptase PCR (RTrtPCR) analysis
  Respiratory specimens will be stored at 2-8 degrees C and processed within 24-48 hours of collection
  Serum and whole blood for immune assays will be processed and then frozen at -20 degrees C or in liquid nitrogen until tested in batch assays
  All blood specimens will be sent to the laboratory for immunologic assays
  Cheek swabs will be used for HLA typing
  Saliva specimens will be used for immunologic assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cincinnati IMPRINT birth cohort: mother-infant pairs enrolled at or after week 34 in pregnancy and followed over three flu seasons, up to four years of age.

SUMMARY:
The primary aim is to define the immune responses to the infant's initial influenza exposure (vaccine or infection) and how that affects the immune response to subsequent influenza exposures

DETAILED DESCRIPTION:
Vaccination is a leading public health intervention for reducing morbidity and mortality from influenza worldwide. Vaccine optimization is hampered by lack of understanding the natural history of infection and immunity, including the full complement of maternal immunity imparted to infants. This gap in understanding can be addressed only through a well-designed birth cohort study. Up to 1500 mother-infant pairs will be enrolled at or after week 34 in pregnancy over three flu seasons, up to four years of age depending on birth month, at two sites. Follow-up will occur from the third trimester until the child is three to four years of age, along with medical records review to ascertain outcomes not captured through weekly illness and respiratory surveillance, and medical record review up to 18 years of age. The primary aim is to rigorously document the natural history of infection and immune response to influenza in study infants for at least three entire flu seasons.

ELIGIBILITY:
Inclusion Criteria:

* Mother pregnant and ≥ 34 weeks gestation and ≥ 18 yrs. of age
* Plans to deliver at local hospital
* Lives within designated home zip codes:
* No plans to move outside study area within study timeframe
* Cell phone that can be used for text messaging
* Singleton live born infant, born ≥ 34 weeks gestational age (GA)

Exclusion Criteria:

* Fetal or infant death prior to maternal hospital discharge
* Mother known to be infected with HIV based on medical records
* Major congenital anomalies, prenatally diagnosed or other major disorder or anomaly as determined by the PI
* Reported use of heroin, cocaine or methamphetamines during pregnancy
* Adoptive infant
* Enrolled in any investigational vaccine trial or other interventional randomized, clinical trial involving the mother or infant that the PI's deem to be in conflict with study outcomes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will seek to obtain a balanced temporal distribution of the cohort births to account for seasonal variations in influenza transmission patterns. We will seek to enroll 30 eligible women per month by posting advertisements via study flyers and brochures in the maternal clinics, social media, institutional wide emails, and each of the enrollment clinic sites. Our staff will screen pregnant women in clinic settings for inclusion/exclusion criteria and then consent and enroll those eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune response to influenza virus infection | 4 years
  Evaluate the immune response to influenza virus infections due to various subtypes in healthy children from birth to 4 years of age in a maternal-infant birth cohort
Immune response to influenza vaccination | 4 years
  Evaluate the immune response to influenza vaccination in healthy children from 6 months to 4 years of age in a maternal-infant birth cohort

CONTACTS AND LOCATIONS:
Overall Officials: Mary Staat, MD,MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No